CLINICAL TRIAL: NCT04160312
Title: Open-labelled, Crossover and Randomized Study With Mitopure™ (Proprietary Urolithin A) Dietary Supplementation Compared to Pomegranate Juice Intake: A Bioavailability Study in Healthy Adults (NOURISH)
Brief Title: Mitopure™ (Proprietary Urolithin A) Bioavailability in Healthy Adults
Acronym: NOURISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AFCRO-110 / 19.01.AMZ
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Healthy; Healthy Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitopure™ (Proprietary Urolithin A) (Experimental): Fruit flavored food sachet containing fixed dose of Mitopure™ (Proprietary Urolithin A)
  Interventions: Dietary Supplement: Mitopure™ (Proprietary Urolithin A)
- Pomegranate Juice (Experimental): 100% Pomegranate juice equivalent to a glass of juice
  Interventions: Dietary Supplement: Pomegranate Juice

INTERVENTIONS:
Dietary Supplement: Mitopure™ (Proprietary Urolithin A) — Fruit flavored sachet containing fixed dose of Mitopure™ (Proprietary Urolithin A)
  Arms: Mitopure™ (Proprietary Urolithin A)
Dietary Supplement: Pomegranate Juice — 100% Pomegranate juice (approximately 1 glass equivalent)
  Arms: Pomegranate Juice

SUMMARY:
This is a single-center, two-period, crossover, randomized, open labelled study enrolling 100 healthy subjects to evaluate the Urolithin A producer status and to compare bioavailabilty of direct dietary supplementation with Mitopure™ (proprietary Urolithin A) to dietary exposure with pomegranate juice

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 to 80 years of age;
2. Is in general good health, as determined by the clinical research team;
3. Willingness to consume investigational product, complete questionnaires and to complete all clinic visits;
4. Have given voluntary, written, informed consent to participant in the study;

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial;
2. Alcohol or drug abuse within the last 6 months;
3. Volunteers who plan to donate blood during the study or within 30 days of completing the study;
4. Subject has a known allergy to the test material's active or inactive ingredients;
5. Subjects with unstable medical conditions;
6. Clinically significant abnormal laboratory results at screening;
7. Participation in a clinical research trial within 30 days prior to randomization;
8. Allergy or sensitivity to study ingredients; lactose intolerance.
9. Individuals who are cognitively impaired and/or who are unable to give informed consent;
10. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.
11. Has taken antibiotics within the previous 30 days;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Absolute change from T0 to T+24 hours in the Urolithin A (UA) group as compared to Pomegranate Juice (PJ) group in UA- glucuronide plasma levels. | 2 days

SECONDARY OUTCOMES:
Absolute change from T0 to T+24 hours in the UA group as compared to PJ group in UA- glucuronide blood spot levels | 2 days
Absolute change from T0 to T+6 hours in the UA group as compared to PJ group in UA- glucuronide plasma levels. | 1 day
Absolute change from T0 to T+6 hours in the UA group as compared to PJ group in UA- glucuronide blood spot levels. | 1 day
Change in AUC from T0 to T+6 and/or T+24 in the UA group as compared to the PJ group in UA glucuronide levels | 2 days
Absolute change from T0 to T6 hours and/or to T24 hours in the UA group as compared to PJ group in UA aglycone (parent) plasma levels | 2 days
Change in AUC from T0 to T+6 and/or T+24 in the UA group as compared to the PJ group in UA aglycone (parent) plasma levels | 2 days
Absolute change from T0 to T6 hours and/or to T24 hours in the UA group as compared to PJ group in UA sulfate plasma levels | 2 days
Change in AUC from T0 to T6 hours and/or to T24 hours in the UA group as compared to PJ group in UA sulfate plasma levels | 2 days
To assess prevalence of UA producers following consumption of fixed volume of Pomegranate juice in a healthy US population | 2 days
Differences between UA producers and non-producers at baseline for Hand grip strength using a calibrated JAMAR® Hydraulic Hand Dynamometer | 2 days
Differences between UA producers and non-producers at baseline for gait speed using the 4-meter gait speed test | 2 days
Differences between UA producers and non-producers at baseline for physical activity levels assessed via the International Physical Activity Questionnaire. | 2 days
  Questionnaire consists of questions that provide information on the physical activity in the last 7 days. Activities include total of duration and frequency from walking, moderate activity and severe physical activity. Accordingly,there are 3 activity levels: Inactive,minimal active and very active.The lowest level of physical activity is inactive and the highest level of physical activity is very active.
Differences between UA producers and non-producers at baseline for energy levels assessed via the Lee-Visual Analogue Scale to assess Fatigue (VAS-F). | 2 days
  The scale consists of 18 items relating to the subjective experience of fatigue. Scores fall between 0 (not fatigued at all) and 100 (extremely fatigued).
Differences between UA producers and non-producers at baseline for gut microbiome. Fecal samples will be used to extract DNA and shotgun sequencing will be performed to assess global microbiome differences at the species level. | 2 days
Differences between UA producers and non-producers at baseline for plasma metabolome. Metabolites in serum will be measured by metabolomic mass spectrometry | 2 days
Differences between UA producers and non-producers at baseline for blood biochemistry metabolic profile as assessed via lipid profile in plasma. | 2 days
Differences in consumer perception on the study investigation food products overall taste using a consumer perception Likert scale | 1 day
  Scale, of 1 to 5 where 1 is dislike extremely and 5 is like extremely

CONTACTS AND LOCATIONS:
Overall Officials: Ali Keshavarzian, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Atlantia Food Clinical Trials CRO (Northwestern University campus), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No